CLINICAL TRIAL: NCT03780972
Title: A Phase 1 Open-Label, Dose Escalation Study to Assess the Safety and Tolerability of Intravitreal ONL1204 in Patients With Macula-off, Rhegmatogenous Retinal Detachment
Brief Title: A Study to Evaluate the Safety and Tolerability of ONL1204 in Patients With Macula-off, Rhegmatogenous Retinal Detachment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ONL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONL1204-RRD-001
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Rhegmatogenous Retinal Detachment - Macula Off
MeSH Terms: interventions — ONL1204; Intravitreal Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Dose A (Active Comparator): Intravitreal injection of 50 μl of ONL1204 liquid formulation to deliver dose 1
  Interventions: Drug: ONL1204; Procedure: Intravitreal Injection; Procedure: Collection of ocular fluids
- Cohort 2 Dose B (Active Comparator): Intravitreal injection of 100 μl of ONL1204 liquid formulation to deliver dose 2
  Interventions: Drug: ONL1204; Procedure: Intravitreal Injection; Procedure: Collection of ocular fluids
- Cohort 3 Dose C (Active Comparator): Intravitreal injection of 50 μl of ONL1204 liquid formulation to deliver dose 3
  Interventions: Drug: ONL1204; Procedure: Intravitreal Injection; Procedure: Collection of ocular fluids
- Cohort 4 Dose D (Active Comparator): Intravitreal injection of 100 μl of ONL1204 liquid formulation to deliver dose 4
  Interventions: Drug: ONL1204; Procedure: Intravitreal Injection; Procedure: Collection of ocular fluids

INTERVENTIONS:
Drug: ONL1204 — Administration of ONL1204 - inhibitor of Fas(CD95) signaling by intravitreal injection
Procedure: Intravitreal Injection — Injection of study drug into the eye
Procedure: Collection of ocular fluids — vitreous and aqueous fluid collection by a tap and during vitrectomy

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ONL1204 in participants with Macula-off, Rhegmatogenous Retinal Detachment (RRD). RRD is an acute and serious vision threatening condition in which a tear in the retina, typically resulting from a vitreous detachment, allows liquid to accumulate under the retina, detaching the photoreceptor (PR) layer of the retina from the retinal pigment epithelium (RPE). As the RPE is the principal source of nutritional support for the PR layer, the photoreceptors begin a cascade of inflammation and cell death. Photoreceptor cell death is the primary mechanism of vision loss after retinal detachment.

ONL1204 is a first-in-class inhibitor of Fragment Apoptosis Stimulator receptor (Fas)-mediated cell death. ONL1204 has demonstrated protection of multiple retinal cell types in numerous preclinical models of acute ocular injury. This will be a first-in-human (FIH) study to evaluate safety and tolerability of a single-dose of ONL1204 in participants with macula-off RRD. The standard of care for surgical repair of macula-off RRD is reattachment surgery within 7 days of the macula detaching. Participants in this study will receive a single intravitreal injection upon diagnosis and enrollment in the study, followed by standard of care surgery. The surgery includes vitrectomy, a procedure that removes the bulk of drug remaining in the vitreous.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ≥ 18 to 80 years old
2. Able to give informed consent and comply with all study visits and procedures
3. Patients who:

   1. Present between 1 week (7 days) and 4 weeks (28 days) of a macula-off RRD (based on patient-reported history of loss of central vision)
   2. For whom standard retinal reattachment surgery by means of a pars plana vitrectomy (with or without scleral buckle) and gas tamponade is indicated, and
   3. In the opinion of the investigator, can safely undergo all study procedures.
4. Best corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity of 20/100 to hand motion in the study eye
5. Best corrected ETDRS visual acuity in the fellow eye of 20/60 or better

Exclusion Criteria:

1. Presence of giant retinal tear defined as greater than 3 clock hours or other type of complex retinal detachment in the study eye
2. Presence of vitreous hemorrhage in the study eye
3. Presence of ocular or periocular infection or intraocular inflammation in either eye
4. Intraocular Pressure > 22 mmHg in the study eye
5. Any other significant ocular disease in the study eye including media opacity that, in the opinion of the investigator, would preclude a visual acuity of at least 20/25 following successful vitrectomy or limit adequate visibility of the retina
6. Any other ocular pathology in the study eye requiring treatment with topical ophthalmic drops or intravitreal injection
7. History of previous ocular surgery in the study eye other than uncomplicated cataract surgery with posterior chamber intraocular lens and intact posterior capsule (which must have occurred at least 6 months prior to the baseline visit)
8. Participation in other clinical trials or use of any other investigational drugs or devices within 3 months prior to study participation
9. Females who are pregnant or lactating and women of childbearing potential who are not using adequate contraceptive precautions (e.g., intrauterine device, oral contraceptives, barrier method, or other contraception deemed adequate by the investigator)
10. Known retinopathy, known hepatic disease (or history of significant chronic liver disease), or known renal disease. Patients with diabetes and no known retinopathy may be enrolled
11. History of uncontrolled hypertension
12. History of stroke, transient ischemic attack, or major cardiac surgery within 3 months prior to study, or current treatment for systemic infection
13. Any ocular or systemic condition that in the opinion of the investigator could compromise the safety of the patient, or may interfere with the safety and tolerability assessments or study procedures of the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Simunovic, M.D., Principal Investigator — Save Sight Institute, Sydney Eye Hospital, Australia
Locations (4):
- Australia (4):
  - Save Sight Institute, Sydney Eye Hospital, Sydney, New South Wales
  - Royal Adelaide, Melbourne, Victoria
  - Queensland Eye Institute, Melbourne, Victoria
  - Center for Eye Rearch Australia, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 Dose A: Intravitreal injection of 50 μl of ONL1204 liquid formulation to deliver dose A
  ONL1204: Administration of ONL1204 - inhibitor of Fas(CD95) signaling by intravitreal injection
  Intravitreal Injection: Injection of study drug into the eye
  Collection of ocular fluids: vitreous and aqueous fluid collection by a tap and during vitrectomy
- Cohort 2 Dose B: Intravitreal injection of 100 μl of ONL1204 liquid formulation to deliver dose B
  ONL1204: Administration of ONL1204 - inhibitor of Fas(CD95) signaling by intravitreal injection
  Intravitreal Injection: Injection of study drug into the eye
  Collection of ocular fluids: vitreous and aqueous fluid collection by a tap and during vitrectomy
- Cohort 3 Dose C: Intravitreal injection of 50 μl of ONL1204 liquid formulation to deliver dose C
  ONL1204: Administration of ONL1204 - inhibitor of Fas(CD95) signaling by intravitreal injection
  Intravitreal Injection: Injection of study drug into the eye
  Collection of ocular fluids: vitreous and aqueous fluid collection by a tap and during vitrectomy
- Cohort 4 Dose D: Intravitreal injection of 100 μl of ONL1204 liquid formulation to deliver dose D
  ONL1204: Administration of ONL1204 - inhibitor of Fas(CD95) signaling by intravitreal injection
  Intravitreal Injection: Injection of study drug into the eye
  Collection of ocular fluids: vitreous and aqueous fluid collection by a tap and during vitrectomy
Period: Overall Study
Arm/Group | Cohort 1 Dose A | Cohort 2 Dose B | Cohort 3 Dose C | Cohort 4 Dose D
Started | 4 | 4 | 4 | 2
Completed | 4 | 4 | 4 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Dose A | Cohort 2 Dose B | Cohort 3 Dose C | Cohort 4 Dose D | Total
Number analyzed (Participants) | 4 | 4 | 4 | 2 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 3 | 0 | 7
  >=65 years | 3 | 1 | 1 | 2 | 7
Age, Continuous [Mean (Full Range); unit: years] | 67.5 [62 to 70] | 54.5 [43 to 68] | 58 [43 to 84] | 67.5 [65 to 70] | 61 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 1 | 3
  Male | 4 | 2 | 4 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 2 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 3 | 4 | 2 | 2 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 4 | 4 | 4 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event (AE) Reporting
Description: AEs restricted to treatment-emergent AEs (TEAEs) only. Ocular and non-ocular AEs reported separately.
  See AE Reporting Table for descriptive ocular and non-ocular AE findings.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Dose A | Cohort 2 Dose B | Cohort 3 Dose C | Cohort 4 Dose D
Number analyzed (Participants) | 4 | 4 | 4 | 2
Participants | 3 | 3 | 3 | 2

2. Primary Outcome: BCVA (LogMAR) at Final Study Visit
Description: BCVA was performed in the study eye using ETDRS methodology and letters read were converted to a logMAR value using the following equation: logMAR = -0.02 × ETDRS + 1.7.
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: logMAR
Arm/Group | Cohort 1 Dose A | Cohort 2 Dose B | Cohort 3 Dose C | Cohort 4 Dose D
Number analyzed (Participants) | 4 | 4 | 4 | 2
logMAR | 0.52 [0.2 to 0.7] | 0.50 [0.2 to 0.8] | 0.77 [0.5 to 1.3] | 0.46 [0.2 to 0.7]

3. Other Pre Specified Outcome: Exploratory Outcome-ONL1204 Concentration
Description: Measurement of ONL1204 in plasma (ng/ml) after drug administration.
  For all subjects, the concentration was <LLOQ.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Cohort 1 Dose A | Cohort 2 Dose B | Cohort 3 Dose C | Cohort 4 Dose D
Number analyzed (Participants) | 4 | 4 | 4 | 2
ng/ml | NA (NA) — All samples collected were below the LLOQ. | NA (NA) — All samples collected were below the LLOQ. | NA (NA) — All samples collected were below the LLOQ. | NA (NA) — All samples collected were below the LLOQ.

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cohort 1 Dose A | Cohort 2 Dose B | Cohort 3 Dose C | Cohort 4 Dose D
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/4 | 2/4 | 0/2
Other Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 3/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Dose A (N=4) | Cohort 2 Dose B (N=4) | Cohort 3 Dose C (N=4) | Cohort 4 Dose D (N=2)
Retinal Re-Detachment (Eye disorders) | 0 (0) | 2 (3) | 2 (3) | 0 (0)
Intraocular Inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Dose A (N=4) | Cohort 2 Dose B (N=4) | Cohort 3 Dose C (N=4) | Cohort 4 Dose D (N=2)
Cataract or Worsening of Cataract (Eye disorders) | 0 | 1 | 2 | 0
Ocular pain post intravitreal injection/injury (Eye disorders) | 1 | 0 | 0 | 0 — Ocular pain post intravitreal injection/injury, poisoning and procedural complications/procedural pain
Elevated Intraocular Pressure (Eye disorders) | 1 | 1 | 0 | 1
Redness/Ocular Hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Nerve Fiber Lesions/OCT Abnormalities (Eye disorders) | 1 | 0 | 0 | 0 — White nerve fibre layer lesions/optical coherence tomography abnormal
Food Poisoning/Gastrointestinal Disorders (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Covid-19 Positive (General disorders) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Redness of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ocular Pain (Eye disorders) | 0 | 1 | 1 | 0
Anterior Uveitis (Eye disorders) | 0 | 2 | 0 | 0
Intraretinal Fluid (Eye disorders) | 0 | 1 | 0 | 0
Ocular Inflammation (Eye disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Pain Frontal Bone Above Left Eye (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Gall Bladder Stones (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abdomen Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Bilateral Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cryo Scars (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Retinal Hole (Eye disorders) | 0 | 0 | 1 | 0
Punctate Epithelial Erosions (Eye disorders) | 0 | 0 | 1 | 0
Floaters (Eye disorders) | 0 | 0 | 1 | 0
Intraocular Lens Opacified (Eye disorders) | 0 | 0 | 1 | 0
Lattice with Atrophic Hole (Eye disorders) | 0 | 0 | 1 | 0
Retinal Degeneration (Eye disorders) | 0 | 0 | 1 | 0
Gel Like Substance in Vitreous Cavity (Eye disorders) | 0 | 0 | 0 | 1
Intraretinal Fluid (Eye disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03780972/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03780972/SAP_001.pdf